CLINICAL TRIAL: NCT00979043
Title: The Arthritis, Diet, and Activity Promotion Trial
Acronym: ADAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00003799; P60AG010484-07 (NIH)
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2023-04-14 (Actual); Status verified 2018-07

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; weight-loss; exercise; obesity; physical function; total mortality
MeSH Terms: conditions — Osteoarthritis, Knee; Weight Loss; Motor Activity; Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dietary weight-loss (Active Comparator): The goal of the dietary weight-loss intervention was to produce and maintain a mean weight-loss of 5% initial body weight during the 18-month intervention, using dietary counseling and behavior modification.
  Interventions: Behavioral: Dietary Weight-loss
- Exercise (Active Comparator): Participants participated in resistance training (15 minutes) and aerobic exercise (30 minutes) 3d/week for 18-months. The first 4-months of the exercise training were facility-based. After 4-months, participants were allowed to transition to a home-based intervention if they chose to.
  Interventions: Behavioral: Exercise
- Dietary weight-loss & exercise (Active Comparator): Participants received both the dietary weight-loss and exercise interventions for 18-months
  Interventions: Behavioral: Dietary Weight-loss; Behavioral: Exercise
- Health lifestyle control (No Intervention): The healthy-lifestyle control served as the usual care comparison group. For 3 months, participants met monthly with a health educator to discuss topics such as osteoarthritis, obesity, and exercise. Regular phone contact was maintained during months 4-18.

INTERVENTIONS:
Behavioral: Dietary Weight-loss — The goal of the dietary weight-loss intervention was to produce and maintain a mean weight-loss of 5% initial body weight during the 18-month intervention, using dietary counseling and behavior modification.
  Arms: Dietary weight-loss; Dietary weight-loss & exercise
Behavioral: Exercise — Participants participated in resistance training (15 minutes) and aerobic exercise (30 minutes) 3d/week for 18-months. The first 4-months of the exercise training were facility-based. After 4-months, participants were allowed to transition to a home-based intervention if they chose to.
  Arms: Dietary weight-loss & exercise; Exercise

SUMMARY:
The primary purpose of this study was to determine the effect of dietary weight-loss, exercise training, or a combination of both on physical function in overweight and obese adults with knee osteoarthritis (OA). In secondary analyses, the effect of weight-loss and/or exercise on OA progression, self-reported pain and inflammation were examined. In post-trial analyses, the effect of dietary weight-loss on total mortality was determined.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years.
* BMI ≥ 28 kg/m2.
* Knee pain on most days of the month.
* Sedentary lifestyle pattern (<20 min exercise per week for last 6 months)
* Self-reported difficulty with at least one of the following: walking 1/4 mile, climbing stairs, kneeling, bending, stooping, shopping, lifting, self-care.
* Radiographic evidence of grade 1-3 knee osteoarthritis.

Exclusion Criteria:

* Serious medical condition that precludes safe participation in exercise such as heart disease (angina, congestive heart failure), severe hypertension, COPD, renal or liver disease, insulin-dependent diabetes.
* Mini-mental state exam score <24.
* Inability to walks without a cane.
* Reported alcohol consumption >14 drinks/week.
* Inability to complete protocol.
* ST segment depression.
* Participation in another research study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 1997-11; Primary Completion 2000-12 (Actual); Study Completion 2000-12 (Actual)

PRIMARY OUTCOMES:
self-reported physical function (WOMAC scale) | baseline, 6-months, 18-months

SECONDARY OUTCOMES:
6-minute walking distance | baseline, 6-months, 18-months
timed stair climbing | baseline, 6-months, 18-months
weight-loss | baseline, 6-months, 18-months
self-reported pain | baseline, 6-months, 18-months
progression of knee osteoarthritis, measured radiographically | baseline, 6-months, 18-months
chronic inflammation, measured according to CRP, IL-6, IL-6 soluble receptor, TNF-alpha, TNF alpha receptors 1 and 2 | baseline and 18-months
total mortality | 7-9 yrs post-trial

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Messier, PhD, Principal Investigator — Wake Forest University
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States

REFERENCES:
- [Result] Messier SP, Loeser RF, Miller GD, Morgan TM, Rejeski WJ, Sevick MA, Ettinger WH Jr, Pahor M, Williamson JD. Exercise and dietary weight loss in overweight and obese older adults with knee osteoarthritis: the Arthritis, Diet, and Activity Promotion Trial. Arthritis Rheum. 2004 May;50(5):1501-10. doi: 10.1002/art.20256. PMID 15146420
- [Result] Nicklas BJ, Ambrosius W, Messier SP, Miller GD, Penninx BW, Loeser RF, Palla S, Bleecker E, Pahor M. Diet-induced weight loss, exercise, and chronic inflammation in older, obese adults: a randomized controlled clinical trial. Am J Clin Nutr. 2004 Apr;79(4):544-51. doi: 10.1093/ajcn/79.4.544. PMID 15051595
- [Result] Miller GD, Nicklas BJ, Davis CC, Ambrosius WT, Loeser RF, Messier SP. Is serum leptin related to physical function and is it modifiable through weight loss and exercise in older adults with knee osteoarthritis? Int J Obes Relat Metab Disord. 2004 Nov;28(11):1383-90. doi: 10.1038/sj.ijo.0802737. PMID 15278105
- [Result] Chua SD Jr, Messier SP, Legault C, Lenz ME, Thonar EJ, Loeser RF. Effect of an exercise and dietary intervention on serum biomarkers in overweight and obese adults with osteoarthritis of the knee. Osteoarthritis Cartilage. 2008 Sep;16(9):1047-53. doi: 10.1016/j.joca.2008.02.002. Epub 2008 Mar 24. PMID 18359648